CLINICAL TRIAL: NCT07153653
Title: Effect of Baduanjin Exercise Intervention on Pregnancy-Related Pain and Quality of Life: A Randomized Controlled Trial
Brief Title: Managing Pregnancy Pain With Baduanjin Exercise
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: K5090
Record Dates: First submitted 2025-07-27; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-03

CONDITIONS: Pregnancy-related Low Back and Pelvic Pain; Pregnancy
Keywords: pregnancy-related Low back and pelvic pain; pregnancy; low back pain; pelvic girdle pain
MeSH Terms: conditions — Pelvic Pain; Low Back Pain; Pelvic Girdle Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baduanjin Group (Experimental): Prenatal Baduanjin Exercise Program
  Interventions: Behavioral: Prenatal Baduanjin Exercise Program
- Standard Clinic Prenatal Care (No Intervention)

INTERVENTIONS:
Behavioral: Prenatal Baduanjin Exercise Program — A structured 12-week program featuring Baduanjin, a traditional Chinese mind-body exercise involving gentle, flowing movements. Participants receive 24 online instructional sessions (approximately 2 s
  Arms: Baduanjin Group

SUMMARY:
This is a randomized controlled trial studying whether a 12-week Baduanjin exercise program (a traditional Chinese mind-body exercise) can reduce low back pain and improve quality of life in pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Single pregnancy (carrying one fetus).
* Gestational age: 14-20 weeks at enrollment.
* No contraindications to exercise during pregnancy (as determined by medical evaluation).

Exclusion Criteria:

* Adverse pregnancy symptoms:
* Dizziness, blurred vision, vaginal bleeding, or other high-risk signs.
* Pre-existing medical conditions: Orthopedic, cardiovascular, or psychiatric diseases; cognitive impairment.
* Pregnancy complications: Preterm labor, placenta previa.
* Inability to attend regular prenatal check-ups.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Low Back Pain Severity | Baseline, 6 weeks, post-intervention (12 weeks)
  Measured using Numerical Rating Scale (NRS) where 0 = no pain and 10 = worst imaginable pain. Assesses self-reported low back/pelvic girdle pain intensity.

SECONDARY OUTCOMES:
Back Disability | Baseline, 6 weeks, post-intervention (12 weeks)
  Functional limitations measured using: Chinese Oswestry Disability Index. Higher scores indicate greater disability.
Pelvic Disability | Baseline, 6 weeks, post-intervention (12 weeks)
  Functional limitations measured using: Pelvic Girdle Questionnaire. Higher scores indicate greater disability.
Urinary Incontinence | Baseline, 6 weeks, post-intervention (12 weeks)
  Measured using: ICIQ-SF (International Consultation on Incontinence Questionnaire-Short Form)). Higher scores indicate worse symptoms/impact.
Urinary Incontinence Severity | Baseline, 6 weeks, post-intervention (12 weeks)
  Measured using: IIQ-7 (Incontinence Impact Questionnaire-7). Higher scores indicate greater disability.

CONTACTS AND LOCATIONS:
Overall Officials: Liangkun Ma, Study Chair — Chinese Academy of Medical Science & Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No